CLINICAL TRIAL: NCT06076148
Title: Aging Well by Being Connected - Phase 1
Brief Title: Virtual Reality and Technologies for Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); SEC Fonds Immobilier Groupe Maurice (Unknown); Fédération Québécoise des Loisirs en Institution (Unknown); Fédération de l'Age D'Or du Québec (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RD-407_VR 50+
Record Dates: First submitted 2023-03-06; First posted 2023-10-10 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Aging Well
Keywords: Aging well; Virtual reality; Immersive technology; Older adults; Physical activity; Cognitive activity; Social behaviour
MeSH Terms: conditions — Motor Activity; Social Behavior

STUDY DESIGN:
Intervention Model Description: All participants will test both multiplayer and individual games. Order of testing is reversed in between arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual then multiplayer games (Experimental): Participants of this group will conduct the sessions in the following order : Focus group about individual virtual reality games then Focus group about multiplayer virtual reality games.
  Interventions: Device: Virtual reality games
- Multiplayer then individual games (Experimental): Participants of this group will conduct the sessions in the following order : Focus group about multiplayer virtual reality games then Focus group about individual virtual reality games.
  Interventions: Device: Virtual reality games

INTERVENTIONS:
Device: Virtual reality games — three individual games (physical, cognitive and relaxation) and two multiplayer games will be tested.

SUMMARY:
The objective of this clinical trial is to understand the determinants and opportunities for acceptance of immersive technologies to support physical, cognitive, and social health and the possibilities for "aging well" among the new generation of older adults. The main questions it aims to answer are:

* What are the needs and expectations in terms of immersive activities and intervention methods according to age?
* Do different game modes influence the needs and expectations in immersive activities of this population? 50 participants will be asked to complete a preliminary questionnaire about their activity habits and preferences. They will then be invited to participate in individual or multiplayer virtual reality game trials, a post-trial discussion about their experience and a questionnaire completion.

ELIGIBILITY:
Inclusion Criteria:

* Be 50 years old or older

Exclusion Criteria:

* Having functional limitations
* Having cognitive impairments
* Being at risk of epilepsy
* Not being autonomus
* Having a pacemaker

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TOPMED, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 candidates were screened for eligibility between April 14, 2023 and May 23, 2023.
Pre-assignment Details: 7 participants were randomized.
Period: Overall Study
Arm/Group | Individual Then Multiplayer Games | Multiplayer Then Individual Games
Started | 5 | 2
Completed | 5 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Then Multiplayer Games | Multiplayer Then Individual Games | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Customized [Count of Participants; unit: Participants]
  Over 50 years old | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 2 | 7
Interest in immersive activities [Mean (Standard Deviation); unit: units on a scale] — Total score for 13 questions with 3 point scale (low, medium, high respectively scored 1,2,3). Minimum=13(low interest); Maximum=39(High interest);
  units on a scale | 30.4 (3.6) | 39 (0) | 32.9 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Perception of Immersive Technologies Experience
Description: 4 open questions were asked during the focus group about satisfaction with the trials. The answers were assessed through a qualitative data theme analysis. The total number of mentionned items by the intervention group is reported for two themes: appreciated items(things that the participants liked during the games), less appreciated items (things that the participants didn't like during the games).
Time Frame: Immediately after each intervention (Week 1, Week 2)
Population: All participants who received the intervention.
Measure: Number; unit: Number of mentionned items
Arm/Group | Individual Then Multiplayer Games | Multiplayer Then Individual Games
Number analyzed (Participants) | 5 | 2
Number of mentionned items
  Appreciated items, week 1 | 24 | 19
  Less appreciated items, week 1 | 7 | 3
  Appreciated items, week 2 | 11 | 23
  Less appreciated items, week 2 | 0 | 4

2. Primary Outcome: Integration of Virtual Reality
Description: 3 open questions were asked during the focus group about intergration of virtual reality(VR) in the daily lives of the participants. The answers were assessed through a qualitative data theme analysis. The total number of mentionned items by the intervention group is reported for two themes: obstacles(factors that make the integration of VR harder in the participant's life), facilitating factors(factors that make the integration of VR easier in the participant's life), .
Time Frame: Immediately after each intervention (Week 1, Week 2)
Population: All participants who received the intervention.
Measure: Number; unit: Total number of mentionned items
Arm/Group | Individual Then Multiplayer Games | Multiplayer Then Individual Games
Number analyzed (Participants) | 5 | 2
Total number of mentionned items
  Obstacles, week 1 | 10 | 12
  Facilitating factors, week 1 | 10 | 5
  Obstacles, week 2 | 7 | 10
  Facilitating factors, week 2 | 0 | 11

3. Primary Outcome: Acceptability of Immersive Technologies
Description: 1 open question was asked during the focus group about intention to use virtual reality(VR) in the daily lives of the participants. The answers were assessed through a qualitative data theme analysis. The total number of mentionned items by the intervention group is reported for one theme: use case of VR items(ways of using VR in the participants daily lives).
Time Frame: Immediately after each intervention (Week 1, Week 2)
Population: All participants who received the intervention.
Measure: Number; unit: Number of mentionned items
Arm/Group | Individual Then Multiplayer Games | Multiplayer Then Individual Games
Number analyzed (Participants) | 5 | 2
Number of mentionned items
  use case of VR items, week 1 | 11 | 10
  use case of VR items, week 2 | 5 | 16

4. Primary Outcome: Change From Baseline in Interest in Immersive Activities
Description: Change from baseline in total score for 13 questions with 3 point scale (low, medium, high respectively scored 1,2,3). Minimum=13(low interest); Maximum=39(High interest);
Time Frame: Baseline and immediately after each intervention (Week 1, Week 2)
Population: All participants who received the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individual Then Multiplayer Games | Multiplayer Then Individual Games
Number analyzed (Participants) | 5 | 2
score on a scale
  Week 1 | 3.00 (3.65) | -1.00 (1.41)
  Week 2 | 3.00 (2.45) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during protocol, which lasted up to 4 weeks, only adverse events which happened during sessions were collected.
Groups:
- Individual Games: Focus group about individual virtual reality games
  Virtual reality games: three individual games (physical, cognitive and relaxation)
- Multiplayer Games: Focus group about multiplayer virtual reality games
  Virtual reality games: two multiplayer games were tested.
Arm/Group | Individual Games | Multiplayer Games
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT06076148/Prot_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT06076148/ICF_001.pdf